CLINICAL TRIAL: NCT03663738
Title: Evaluation of the Impact of a Mobile Health App to Improve Self-control and Health Outcomes of Patients With Type 2 Diabetes Mellitus: Pilot Study "NOVAME"
Brief Title: Impact Evaluation of a Mobile Health App to Improve Self-control and Health Outcomes of Patients With Type 2 Diabetes Mellitus (T2DM): Pilot Study "NOVAME"
Acronym: NOVAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Servicio Canario de Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PIFUN32/17
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Masking Description: Researchers who recruited participants and applied the baseline and 3-month questionnaires were not blinded to the allocation sequence. Given the nature of the intervention patients could not be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- health mobile app for T2DM patients (Active Comparator): It consists of a mobile app that will be provided to patients during a period of 12 months, the patient can also continue with the usual care. The application will be synchronized with a server where all the information is recorded for further analysis. The central focus of the application consists of continuous support and monitoring through the app that has a personalized and dynamic virtual coach that will help the patient to adopt healthy habits and change their behaviors through training plans in different areas: exercise physical, healthy eating, therapeutic education and emotional management
  Interventions: Behavioral: mobile app NOVAME
- Control (No Intervention): Receives the usual care as established in the Canary Islands Atherosclerotic Vascular Disease Prevention and Control Program (EVA)

INTERVENTIONS:
Behavioral: mobile app NOVAME — The training program is divided into 3 periods of 21 days, where each day the patient receives a new formation pill. At the end of one of these periods there will be a week of review in which the patient will receive reminders of the contents that he has already received. These pills will help the patient to acquire healthy lifestyle habits and improve the control of the disease. The length of the program is 84 days, and once completed, the patient can repeat or intensify efforts in the areas he considers and continue to have access to the virtual coach. Patients assigned to the intervention group will receive a brief structured explanation on how to use the application and its contents.
  Arms: health mobile app for T2DM patients

SUMMARY:
The objective of this project is to evaluate the effectiveness and cost effectiveness of a health app (NOVAME) designed to improve the self-control of patients with T2DM and their health outcomes. The central focus of NOVAME is the continuous support to the patient and monitoring through the app that will act as a personalized and dynamic virtual coach that will help the patient to adopt healthy habits and change their behaviors through training plans in different areas: exercise physical, healthy eating, therapeutic education and emotional management The design of the evaluation is the randomized clinical trial, in the intervention arm patients will use the app NOVAME and in the control group, patients don't receive any additional educational or supporting activities beyond the usual activities provided by the Canary Islands Health Service (CIHS). The main outcome measure is the change in HbA1c at 3 months, requiring a total of 197 patients to detect a difference of at least 0.4% considering a 10% loss. As secondary measures HbA1c is collected at 12 months and other biochemical results (lipids and glucose), BMI and a series of questionnaires to measure changes in life habits (diet, physical activity), anxiety and depression, knowledge about their disease , degree of empowerment, satisfaction and usability of the app, .. Will be collected at 3 and 12 months. The differences between the arms will be measured with mixed generalized linear models. The cost effectiveness will be calculated by calculating life years adjusted for quality (QALY) and the cost of the disease, including the use of resources reported by patients. The benefits of the technology will be expressed in terms of HbA1c and QALY.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with T2DM diagnosed at least one year prior to study enrolment
2. 18-65 years of age
3. Formal consent to participate in the study
4. Regular use of mobile phone

Exclusion Criteria:

1. Chronic kidney disease≥stage 3b, as defined by the National Kidney Foundation's Kidney Disease Outcomes and Quality Improvement Initiative (KDOQI); urinary albumin to creatinine ratio (UACR) ≥ 300 mg/g and/or urinary protein excretion ≥ 300 mg/24 hours.
2. Acute coronary syndrome (documented angina or myocardial infarction) or stroke in the last six months or class III or IV heart failure, according to the New York Heart Association (NYHA).
3. Proliferative diabetic retinopathy or clinically significant diabetic macular edema requiring previous treatment with retinal photocoagulation, vitrectomy, or intravitreal injections of antivascular endothelial growth factor or triamcinolone acetonide 6 months prior to study inclusion.
4. Uncorrected severe hearing or visual impairment; or corrected visual acuity ≤ 20/40 by any cause.
5. Diabetic foot with ulcers ≥ 2 according to Wagner scale.
6. Liver cirrhosis
7. Cancer unless disease free five years after diagnosis
8. Other terminal illnesses
9. Intellectual retardation, dementia, psychotic diseases.
10. Active substance abuse, alcohol or drugs (must be sober for one year)
11. Pregnancy
12. Insufficient (Spanish) language skills
13. Physical disability limiting participation in group education activities
14. Concurrent participation in another clinical trial or any other investigational study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
HbA1c | Baseline, 3 months, 12 months
  glycosylated hemoglobin

SECONDARY OUTCOMES:
Total cholesterol and its fractions (LDL, HDL and nonHDL), and triglycerides | Baseline, 3 months, 12 months
  triglycerides, Total Cholesterol, LDL Cholesterol, HDL Cholesterol
Glucose | Baseline, 3 months, 12 months
  glucose level
BMI | Baseline, 3 months, 12 months
  Body mass index
Quality of life related to health | Baseline, 3 months, 12 months
  EQ-5D-5L questionnaire. The EQ-5D is a generic instrument of HRQL measurement where the individual assesses their state of health, first in levels of severity by dimensions (descriptive system) and then in a visual analogue scale (VAS) of more general evaluation. The index ranges between the value 1 (best health status) and 0 (death), although there are negative values for the index, corresponding to health status that are valued as worse than death.

CONTACTS AND LOCATIONS:
Locations (1):
- Servicio de Evaluación. Servicio Canario de Salud, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No